CLINICAL TRIAL: NCT06348797
Title: Phase I Clinical Study on Safety and Feasibility of DLL3 Targeted α-PD-L1/4-1BB Modifying Chimeric Antigen Receptor T-cells in Patients With Relapsed or Refractory Small Cell Lung Cancer (SCLC)
Brief Title: Phase I Clinical Study of α-PD-L1/DLL3 CAR-T in Patients With R/R SCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Collaborators: Chengdu Brilliant Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Cancer, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHP01-01
Record Dates: First submitted 2024-03-18; First posted 2024-04-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: Extensive Stage-SCLC; DLL3 CAR-T; Bridge Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- α-PD-L1/4-1BB DLL3 CAR-T (BHP01) Treatment (Experimental): The Patients enrolled will be sequentially assigned to the corresponding dose level, BHP01 was administered intravenous infusion at different cell dose levels. The patients were received multiple-dose infusion according to investigator's evaluation.
  Interventions: Drug: α-PD-L1/4-1BB DLL3 CAR-T (BHP01)

INTERVENTIONS:
Drug: α-PD-L1/4-1BB DLL3 CAR-T (BHP01) — Preconditioning with fludarabine, cyclophosphamide, based chemotherapy regimen at sub-clinical doses; Bridge radiotherapy with 15 Gray (Gy)/5 fractions; α-PD-L1/4-1BB DLL3 CAR-T (BHP01): the first dose was 5x10^5/kg.
  Other Names: Bridge radiotherapy

SUMMARY:
A study to evaluate the safety and feasibility of α-PD-L1/4-1BB DLL3 Chimeric Antigen Receptor (CAR)-T (BHP01) in patients with Relapsed/Refractory Small Cell Lung Cancer (SCLC) and determine the appropriate CAR-T cell dose. Next, In dose expansion phase, patients were assign two groups with/without bridge radiotherapy.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) accounts for about 15% of lung cancers, and two-thirds of cases are metastatic at the time of diagnosis. The inhibitory notch ligand delta-like ligand 3 (DLL3) is aberrantly expressed on the surface of up to 85% of SCLC cells and minimally expressed in normal tissues, making it a compelling therapeutic target. This is a phase I, first-in-human, 3+3 dose escalation study to evaluate the safety and feasibility of BHP01 in patents with relapsed/refractory SCLC who progressed after at least 1 platinum based chemotherapy regimen.This is a dose escalation and dose expansion study. 12-21 patients with relapsed/refractory SCLC are planned to be enrolled (Group Pre-A/A/B/C). After the Dose-limiting toxicity (DLT) observation period of the related dose group finished.16 patients are planned to enroll in dose expansion phase who was assign two groups with/without bridge radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent or refractory small cell lung cancer (SCLC) confirmed by histology or cytology who have relapsed or progressed after treatment with one previous platinum-based regimen;
* Patients can provide sufficient tumor tissue (fresh or paraffin sections, etc.);
* Age 18 ~70 (including boundary), for both men and women;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Life expectancy ≥3 months;
* At least one extracranial measurable lesion (RECIST v1.1) exists；for lesion after radiotherapy， must be confirmed that the lesion has progressed ;
* Patients in limited-stage at the initial diagnosis must undergo radical thoracic radiotherapy and the time of tumor progression is not less than 3 months from the end of radiotherapy, or radical thoracic dose radiotherapy cannot be performed for specific reasons;
* The test results of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C and syphilis were negative at screening;
* Female patients or male reproductive age patients and their partners should agree to effective contraception from sighing Informed Consent Form (ICF) to 6 months after the last BHP01 infusion.

Exclusion Criteria:

* Patients with known primary Central Nervous System (CNS) tumor, or meningeal metastasis, or patients with unstable CNS metastasis (symptomatic, requiring hormonal therapy within 4 weeks before investigational treatment, or no radiographic evidence of stabilization of the lesion for more than 4 weeks);
* Received major surgical procedures （except for diagnosis） within 4 weeks before PBMCs collection, or are expected to require major surgical procedures during the study;
* Received Chinese herbal medicine or Chinese patent medicine for anti-tumor indications within 7 days before Peripheral Blood Mononuclear Cells (PBMCs) collection;
* Patients with a history of idiopathic pulmonary fibrosis, mechanical pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia or idiopathic pneumonia, or evidence of active pneumonia by chest computer tomography (CT) at screening [a history of radiation pneumonia (fibrosis) in the irradiated field may participate in this study];
* Poorly controlled pleural effusion, pericardial effusion, or ascites requiring repeated drainage procedures (once a month or more frequently);
* Poorly controlled or symptomatic hypercalcemia (ionic calcium> 1.5 mmol/L, calcium> 12 mg/dL or corrected calcium> ULN);
* Presence of active or previous autoimmune diseases or immunodeficiencies, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, etc.;
* Severe infection within 4 weeks before the start of PBMCs collection, including but not limited to hospitalization due to infection, bacteremia, severe pneumonia, or any active infection that may affect the patient's safety;
* Serious cardiovascular and cerebrovascular diseases (such as heart disease ≥New York Heart Association class II, myocardial infarction or cerebrovascular accident), unstable arrhythmia or unstable angina pectoris within 3 months before PBMCs collection;
* Previous treatment with DLL 3 target drugs or CAR-T or other gene-modified T cells;
* Received any other Investigational drug within 28 days prior to PBMCs collection;
* A history of mental illness;
* Incapacitated persons or persons with limited capacity;
* pregnant or lactating females; Males or females who are unwilling to use adequate contraception; Females of childbearing potential are required to undergo a pregnancy study during the screening period;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | day1-day28
  Safety

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 year after the enrollment
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1. In the event of PR or CR, the subjects should confirm it no less than 4 weeks after the first evaluation.
Progression-free survival (PFS) | up to 1 year after the enrollment
  The time from CAR-T administration to disease progression or death.
Disease control rate (DCR) | up to 1 year after the enrollment
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%).
Duration of response (DOR) | up to 1 year after the enrollment
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause
Overall-Survival (OS) | up to 1 year after the enrollment
  The period from the first infusion to any cause of death
CAR-T cell numbers | up to 1 year after the enrollment
  Monitoring CAR-T cell numbers in blood to determine the persistence of CAR-T.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn MJ, Cho BC, Felip E, Korantzis I, Ohashi K, Majem M, Juan-Vidal O, Handzhiev S, Izumi H, Lee JS, Dziadziuszko R, Wolf J, Blackhall F, Reck M, Bustamante Alvarez J, Hummel HD, Dingemans AC, Sands J, Akamatsu H, Owonikoko TK, Ramalingam SS, Borghaei H, Johnson ML, Huang S, Mukherjee S, Minocha M, Jiang T, Martinez P, Anderson ES, Paz-Ares L; DeLLphi-301 Investigators. Tarlatamab for Patients with Previously Treated Small-Cell Lung Cancer. N Engl J Med. 2023 Nov 30;389(22):2063-2075. doi: 10.1056/NEJMoa2307980. Epub 2023 Oct 20. PMID 37861218
- [Background] Paz-Ares L, Champiat S, Lai WV, Izumi H, Govindan R, Boyer M, Hummel HD, Borghaei H, Johnson ML, Steeghs N, Blackhall F, Dowlati A, Reguart N, Yoshida T, He K, Gadgeel SM, Felip E, Zhang Y, Pati A, Minocha M, Mukherjee S, Goldrick A, Nagorsen D, Hashemi Sadraei N, Owonikoko TK. Tarlatamab, a First-in-Class DLL3-Targeted Bispecific T-Cell Engager, in Recurrent Small-Cell Lung Cancer: An Open-Label, Phase I Study. J Clin Oncol. 2023 Jun 1;41(16):2893-2903. doi: 10.1200/JCO.22.02823. Epub 2023 Jan 23. PMID 36689692
- [Background] Megyesfalvi Z, Gay CM, Popper H, Pirker R, Ostoros G, Heeke S, Lang C, Hoetzenecker K, Schwendenwein A, Boettiger K, Bunn PA Jr, Renyi-Vamos F, Schelch K, Prosch H, Byers LA, Hirsch FR, Dome B. Clinical insights into small cell lung cancer: Tumor heterogeneity, diagnosis, therapy, and future directions. CA Cancer J Clin. 2023 Nov-Dec;73(6):620-652. doi: 10.3322/caac.21785. Epub 2023 Jun 17. PMID 37329269
- [Background] Rojo F, Corassa M, Mavroudis D, Oz AB, Biesma B, Brcic L, Pauwels P, Sailer V, Gosney J, Miljkovic D, Hader C, Wu M, Almarez T, Penault-Llorca F. International real-world study of DLL3 expression in patients with small cell lung cancer. Lung Cancer. 2020 Sep;147:237-243. doi: 10.1016/j.lungcan.2020.07.026. Epub 2020 Jul 27. PMID 32745892
- [Background] Jaspers JE, Khan JF, Godfrey WD, Lopez AV, Ciampricotti M, Rudin CM, Brentjens RJ. IL-18-secreting CAR T cells targeting DLL3 are highly effective in small cell lung cancer models. J Clin Invest. 2023 May 1;133(9):e166028. doi: 10.1172/JCI166028. PMID 36951942
- [Background] Zhang Y, Tacheva-Grigorova SK, Sutton J, Melton Z, Mak YSL, Lay C, Smith BA, Sai T, Van Blarcom T, Sasu BJ, Panowski SH. Allogeneic CAR T Cells Targeting DLL3 Are Efficacious and Safe in Preclinical Models of Small Cell Lung Cancer. Clin Cancer Res. 2023 Mar 1;29(5):971-985. doi: 10.1158/1078-0432.CCR-22-2293. PMID 36692420
- [Background] Zhou D, Byers LA, Sable B, Smit MD, Sadraei NH, Dutta S, Upreti VV. Clinical Pharmacology Profile of AMG 119, the First Chimeric Antigen Receptor T (CAR-T) Cell Therapy Targeting Delta-Like Ligand 3 (DLL3), in Patients with Relapsed/Refractory Small Cell Lung Cancer (SCLC). J Clin Pharmacol. 2024 Mar;64(3):362-370. doi: 10.1002/jcph.2346. Epub 2023 Oct 2. PMID 37694295
- [Background] Owen DH, Giffin MJ, Bailis JM, Smit MD, Carbone DP, He K. DLL3: an emerging target in small cell lung cancer. J Hematol Oncol. 2019 Jun 18;12(1):61. doi: 10.1186/s13045-019-0745-2. PMID 31215500